CLINICAL TRIAL: NCT06942104
Title: Imaging of Solid Tumors Using 18F-TRX
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rahul Aggarwal (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Rahul Aggarwal, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 249214; NCI-2025-02615 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor; Solid Carcinoma; Castration-Resistant Prostate Carcinoma; Locally Advanced Clear Cell Renal Cell Carcinoma; Metastatic Clear Cell Renal Cell Carcinoma; Metastatic Malignant Solid Neoplasm; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8; Glioma, Malignant
Keywords: Imaging Studies
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Neoplasm Metastasis; Carcinoma, Renal Cell; Prostatic Neoplasms; Glioma | interventions — Magnetic Resonance Spectroscopy; Biopsy; Blood Specimen Collection; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Diagnostic (18F-TRX) (Experimental): Participants with any solid tumor malignancy with at least 3 metastatic lesions on conventional imaging will receive multiple scans lasting 220 minutes after injection. Participants undergo blood sample collection and may undergo tumor biopsy during screening
  Interventions: Drug: 18F-TRX; Procedure: Positron Emission Tomography (PET)/Computerized tomography (CT); Procedure: Tumor Biopsy; Procedure: Blood Specimen Collection
- Cohort 2: Diagnostic (18F-TRX) (Experimental): Participants with WHO grade 3 or 4 glioma, locally advanced or metastatic clear cell renal cell carcinoma with at least three metastatic lesions on conventional imaging, or metastatic castration-resistant prostate cancer with at least one metastatic lesion on conventional imaging including cross-sectional imaging of the chest, abdomen and pelvis and whole body bone scan or prostate-specific membrane antigen (PSMA) PET scan (n = 30) will receive a single scan lasting 55-144 minutes after injection. Participants may undergo tumor biopsy during screening
  Interventions: Drug: 18F-TRX; Procedure: Positron Emission Tomography (PET)/Computerized tomography (CT); Procedure: Tumor Biopsy

INTERVENTIONS:
Drug: 18F-TRX — Given Intravenously (IV)
  Other Names: Fluorine F 18 TRX
Procedure: Positron Emission Tomography (PET)/Computerized tomography (CT) — Imaging procedure
  Other Names: PET/CT
Procedure: Tumor Biopsy — May undergo tumor biopsy
  Other Names: Biopsy
Procedure: Blood Specimen Collection — Undergo blood sample collection
  Other Names: Blood Sample; Sample Collection
  Arms: Cohort 1: Diagnostic (18F-TRX)

SUMMARY:
This phase I trial tests the safety and effectiveness of 18F-TRX in detecting tumors (cancer) patients with solid tumors. 18F-TRX is an imaging tracer that is used to visualize tumors using a PET scan. It specifically targets and detects labile (unstable) iron levels within tissues, including tumors. Diagnostic procedures, such as 18F-TRX PET/CT or PET/MRI, may help detect tumors in patients with solid tumors

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety of fluorine F 18 trioxolane (18F-TRX) in participants with any solid tumor malignancy with at least 3 metastatic lesions on conventional imaging (Cohort 1); or known or presumed high grade glioma, locally advanced metastatic clear cell renal cell carcinoma with at least 3 lesions on conventional imaging, and metastatic castration-resistant prostate cancer (mCRPC) with at least 1 metastatic lesion on conventional imaging (Cohort 2).

SECONDARY OBJECTIVES:

I. To determine the organ dosimetry and pharmacokinetics of 18F-TRX (Cohort 1).

II. To determine the sensitivity for detection of malignant lesions with 18F-TRX PET in participants with metastatic castration-resistant prostate cancer (n = 30), locally advanced or metastatic clear cell renal cell carcinoma (n = 10), and World Health Organization (WHO) grade 3 or 4 glioma (n = 10) (Cohort 2).

III. To determine the feasibility of lesion detection using 18F-TRX in participants with known or presumed high grade glioma, locally advanced metastatic clear cell renal cell carcinoma with at least 3 lesions on conventional imaging, and mCRPC with at least 1 metastatic lesion on conventional imaging (Cohort 2).

EXPLORATORY OBJECTIVE:

I. To correlate 18F-TRX uptake with Six-Transmembrane Epithelial Antigen of Prostate 3 (STEAP3) expression determined by immunohistochemistry (IHC) evaluation of tumor tissue obtained within 3 months of PET.

OUTLINE:

Participants are assigned to 1 of 2 cohorts:

COHORT 1: Participants receive 18F-TRX intravenously (IV) and undergo up to 8 PET/CT or PET/MRI scans.

COHORT 2: Participants receive 18F-TRX IV and undergo a single scan.

After completion of study intervention, patients are followed up 1-7 days post-injection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Advanced solid tumor malignancy in one of the following cohorts:

  * Cohort 1 (n = 6): Any solid tumor malignancy with at least 3 metastatic lesions on conventional imaging
  * Cohort 2 (n = 50):

    * WHO grade 3 or 4 glioma - patients with known (by integrated molecular and histopathologic diagnosis) or presumed (by imaging; e.g., enhancing necrotic and/or hypervascular intrinsic brain tumor) high grade (WHO grade 3 or 4) glioma (n = 10), Locally advanced or metastatic clear cell renal cell carcinoma with at least three metastatic lesions on conventional imaging (n = 10).
    * Metastatic castration-resistant prostate cancer with at least one metastatic lesion on conventional imaging including cross-sectional imaging of the chest, abdomen and pelvis and whole body bone scan or prostate-specific membrane antigen (PSMA) PET scan (n = 30).
* Ability to understand and the willingness to sign a written informed consent document.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Negative serum or urine pregnancy test (women of childbearing potential only) within 72 hours of baseline procedures.
* Absolute neutrophil count > 1.5 x 10^6/L.
* Platelets > 75,000 x 10^6/L.
* Hemoglobin > 8 g/dL.
* Total bilirubin < 1.5 x upper limit of normal.
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase (SGOT)) < 2.5 x upper limit of normal (< 5 x upper limit of normal in patients with liver metastases on conventional imaging).
* Alanine aminotransferase (ALT)(serum glutamic-pyruvic transaminase (SGPT)) < 2.5 x upper limit of normal (< 5 x upper limit of normal in patients with liver metastases on conventional imaging).
* Creatinine clearance > 50 ml/min, calculated using the Cockcroft-Gault equation.

Exclusion Criteria:

* Individuals with any condition or social circumstance that, in the opinion of the investigator, would impair the participant's ability to comply with study procedures.
* Individuals receiving strong inhibitors or inducers of CYP3A4.
* Uncontrolled active infection or other medical condition that would preclude safe participation in the study as judged by the Investigator.
* Individuals who are pregnant.

  * Individuals of childbearing potential (defined below) must agree to undergo a urine pregnancy test prior to participating in the study scans. Pregnant individuals are excluded because there is an unknown but potential risk for adverse effects in the unborn child secondary to administration of 18F-TRX to the study participant.
  * A female is considered to not be of childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice), if the participant meets either of the following two criteria: (1) has reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause); or (2) has undergone surgical sterilization (i.e., hysterectomy and/or bilateral oophorectomy for removal of uterus and/or ovaries).
* Individuals who are breastfeeding/chestfeeding.

  * Breastfeeding/chestfeeding individuals are excluded because there is an unknown but potential risk for adverse effects in the unborn/nursing child secondary to administration of 18F-TRX to the study participant.
  * Breastfeeding/chestfeeding should be discontinued before administration of 18F-TRX.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment-emergent adverse events | Up to 7 days
  The proportion of participants with any treatment-emergent adverse events will be reported by grade and frequency per the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. All participants who receive the radiotracer injection will be evaluable.

SECONDARY OUTCOMES:
Median Target to Background Ratio (TBR) (Cohort 1) | Day of scan, 1 day
  The measured target-to-background ratios (TBRs) will be reported as the median and range similar to previously reported. The scan time point generating the highest mean TBR will be chosen for subsequent imaging in cohort 2.
Mean radiation-absorbed doses (Cohort 1) | Day of scan, 1 day
  The results from the scans for all patients enrolled will be combined to allow the calculation of mean, standard deviation (SD), and range of radiation-absorbed doses to individual organs as well as effective dose
Sensitivity of tumor lesion detection (Cohort 2) | Day of scan, 1 day
  Sensitivity is the probability that a test will indicate a lesion among those with disease: Sensitivity = True Positive / (True Positive + False Negative). The lesion is defined as positive if the short axis dimension of lymph nodes is greater than 1.5 cm, and organ metastases measure > 1 cm in long axis by conventional imaging. The sensitivity will be obtained by point estimation and 95% confidence interval assuming all lesions are independent to determine the number of tru
Number of lesions detected by fludeoxyglucose F-18 (18F)-TRX positron emission tomography (PET) (Cohort 2) | Day of scan, 1 day
  Number of lesions detected by 18F-TRX PET, but not detected on conventional imaging.
Proportion of patients with one or more metastatic lesion (Cohort 2) | Day of scan, 1 day
  Feasibility will be assessed by conventional imaging (computed tomography and magnetic resonance imaging) and whole-body bone scan, and will be reviewed in conjunction with the 18F-TRX PET images. Conventional imaging will be interpreted as positive by each lesion if the short axis dimension of lymph nodes is greater than 1.5 cm, and organ metastases measure greater than 1 cm in long axis. The gold standard will be conventional imaging. Will be descriptively reported with point estimation and 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No